CLINICAL TRIAL: NCT05863962
Title: Comparative Effects of Jacobson's Relaxation Techniques and Stretching Exercises on Blood Pressure and Anxiety in Preeclampsia
Brief Title: Comparative Effects of Jacobson's Relaxation Techniques and Stretching Exercises in Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0504
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Pre-Eclampsia; Complicating Pregnancy
Keywords: Pregnancy Toxemia,; Muscle Stretching Exercise; High Blood Pressure
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Hypertension | interventions — Walking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching Exercises (Experimental): walking with stretching exercises
  Interventions: Other: walking and Stretching
- Jacobson's Technique (Active Comparator): walking with Jacobson's Relaxation Technique.
  Interventions: Other: walking and Jacobsons relaxation technique

INTERVENTIONS:
Other: walking and Stretching — Stretching exercise will be given for 6 weeks (3 sessions per week). 15 minutes of moderate walking with stretching exercises 5 times a week with Warm up and Cool down. Videos will be provided to participants to follow at home. Participants will be provided forms for home to fill after every session completed and frequency of each exercise
  Arms: Stretching Exercises
Other: walking and Jacobsons relaxation technique — Jacobson's Relaxation Technique will be given for 6 weeks. 15 minutes of moderate walking with Jacobson's Relaxation Technique. Videos will be provided to participants to follow at home. Participants will be provided forms for home to fill after every session completed. Participants will also bring their Pedometer
  Arms: Jacobson's Technique

SUMMARY:
To compare the effect of Jacobson's Relaxation Techniques and stretching exercises on Preeclampsia in pregnant women.

DETAILED DESCRIPTION:
The effectiveness of Jacobson's progressive muscle relaxation technique on maternal, fetal, and neonatal outcomes in women with non-severe preeclampsiain have been studied in an RCT study. Pregnant women who use this technique experience reduced muscle tension and a sense of calm. in one of the study The Effect of Relaxation Techniques on Blood Pressure and Stress Among Pregnant Women with Mild Pregnancy Induced Hypertension were investigated in which Women with mild pregnancy-induced hypertension who used relaxation techniques saw significant improvements in their knowledge, physiological parameters, and blood pressure as well as a reduction in stress.

To the best of the researcher's knowledge, no comparative study has been done to yet to evaluate the efficacy of relaxation and stretching exercise. There is not enough data to determine whether Jacobson's relaxation techniques and stretching exercise reduce preeclampsia in pregnant women. As a result, this study will contribute to the expanding body of knowledge about which approach should be used as an alternative if results from other procedures are comparable

ELIGIBILITY:
Inclusion Criteria:

* Gestational age was exceeding 24 weeks
* BP more than or up to 140/90
* Diagnosed with gestational Hypertension
* Primiparous

Exclusion Criteria:

* Women with history of preterm labor or repeated abortion
* Bleeding
* Intra uterine fetal growth anomalies
* Underlying mental (depression with severe anxiety)
* Cardio respiratory diseases

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Mercury sphygmomanomete | 4 Weeks
  patient have systolic blood pressure of 140 mm Hg or higher and/or a diastolic blood pressure of 90 mm Hg or higher.

SECONDARY OUTCOMES:
Pregnancy related anxiety questionnaire | 4 Weeks
  The degree of anxiety was estimated using Pregnancy related anxiety Questionnaire assessing the symptoms on scale 1 to 5 . 1 being not relevant and 5 relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rana S, Lemoine E, Granger JP, Karumanchi SA. Preeclampsia: Pathophysiology, Challenges, and Perspectives. Circ Res. 2019 Mar 29;124(7):1094-1112. doi: 10.1161/CIRCRESAHA.118.313276. PMID 30920918
- [Background] Pacheco-Romero, J., Introduction to the Preeclampsia. Revista Peruana de Ginecología y Obstetricia, 2017. 63(2): p. 199-206.
- [Background] Nirupama R, Divyashree S, Janhavi P, Muthukumar SP, Ravindra PV. Preeclampsia: Pathophysiology and management. J Gynecol Obstet Hum Reprod. 2021 Feb;50(2):101975. doi: 10.1016/j.jogoh.2020.101975. Epub 2020 Nov 7. PMID 33171282
- [Background] Awad MA, Hasanin ME, Taha MM, Gabr AA. Effect of stretching exercises versus autogenic training on preeclampsia. J Exerc Rehabil. 2019 Feb 25;15(1):109-113. doi: 10.12965/jer.1836524.262. eCollection 2019 Feb. PMID 30899745
- [Background] Ghorbannejad S, MehdizadehTourzani Z, Kabir K, MansourehYazdkhasti. The effectiveness of Jacobson's progressive muscle relaxation technique on maternal, fetal and neonatal outcomes in women with non-severe preeclampsia: a randomized clinical trial. Heliyon. 2022 Jun 13;8(6):e09709. doi: 10.1016/j.heliyon.2022.e09709. eCollection 2022 Jun. PMID 35761936
- [Background] Naseh, Z., P. Bahadoran, and M. Valiani, Effect of Relaxation Technique on Anxiety, Stress, and Depression Scores of High-risk Pregnant Women Prone to Preeclampsia and the Physiological Indicators of Their Babies. Avicenna Journal of Nursing and Midwifery Care, 2022. 30(3): p. 211-220.
- [Background] Abd El Aliem, R.S., E.M. Abd-Elhakam, and S.A. Mustafa, Effect of Self Independence Physical Stretching Exercise on Feto-maternal Outcomes among Mild Preeclamptic Pregnant Women.
- [Background] Vicente Bertagnolli T, Souza Rangel Machado M, Ferreira CJH, Machado JSR, Duarte G, Cavalli RC. Safety of a physical therapy protocol for women with preeclampsia: a randomized controlled feasibility trial. Hypertens Pregnancy. 2018 May;37(2):59-67. doi: 10.1080/10641955.2018.1439059. Epub 2018 Mar 1. PMID 29495906
- [Background] Caughey, M.C., et al., Abstract P035: Feasibility of Stretching Exercise for Prevention of Late-Onset Preeclampsia: A Pilot Trial. Circulation, 2018. 137(suppl_1): p. AP035-AP035.
- [Background] Soliman, G.H., S.M.A. Elalem, and S.M. Elhomosy, The effect of relaxation techniques on blood pressure and stress among pregnant women with mild pregnancy induced hypertension. Asian Journal of Nursing Education and Research, 2017. 7(3): p. 321-329.